CLINICAL TRIAL: NCT02242968
Title: Screening of Volunteers for Clinical Trials of Investigational or Licensed Vaccines or Antiviral Products
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140194; 14-I-0194
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Vaccines; Antiviral Agents; Immunologic Factors; Physiological Effects of Drugs; Anti-Infective Agents
Keywords: Licensed Vaccines; Blood Draw; Investigational Vaccines; Healthy Volunteers; Eligibility Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Male and Female healthy volunteers between aged 18 and 65 years.

SUMMARY:
Background:

- Vaccines and antiviral therapies help prevent and treat diseases. Researchers need a group of healthy volunteers for clinical trials. Clinical trials are studies that test these vaccines and therapies in people.

Objective:

- To screen volunteers for clinical trials for investigational or licensed vaccines or drugs to treat or prevent virus infections.

Eligibility:

- Healthy adults age 18 or older.

Design:

* Participants will be asked questions about their health history, including sexual activity and drug use. They will give blood samples. They may have a physical exam. They may give a urine sample.
* Participants may have the inside of their nose either swabbed or washed with some fluid. The fluid will be collected. They may give a stool sample.
* Participants may have an electrocardiogram. Soft, sticky patches will be attached to participants chest, arms, and legs. They will lie still on a table while the patches detect the heart s electrical signals. A machine will record these signals.
* Participants may have lung function tests. These tests measure the volume of air moving in and out of the lungs. Participants will forcibly blow air into a machine.
* Participants will be told if any tests show a medical problem.
* If a participant is eligible and decides to join an investigational clinical trial, researchers will explain the study and the risks involved. Participants will sign a separate consent for that clinical trial.

DETAILED DESCRIPTION:
Vaccines and antiviral therapies are critical for prevention and treatment of viral diseases. Among other things, testing of vaccines or antiviral medications requires knowing whether the prospective subject has been previously infected by the virus to be studied. We will recruit healthy persons for this study and screen them for their eligibility to potentially participate in clinical trials of investigational or licensed vaccines or antiviral products. In most cases this will involve a medical history, physical examination, and obtaining blood to test for past exposure to one or more viruses being studied in ongoing and upcoming vaccine or antiviral therapy trials. In some cases, blood may be tested for viral DNA or RNA and urine, stool, nasal swab, or nasal wash may be tested for viruses. Additional testing, such as an electrocardiogram (EKG) and pulmonary function tests (PFTs) may also be done. In a subset of volunteers not screening for enrollment in a clinical trial but willing to donate a small volume of blood, nasal swab, throat swab, and/or urine in support of research assay development, no additional testing is anticipated. Overall, this study should 1) help us to identify a group of healthy volunteers who will be eligible, based on testing for their prior exposure to viruses, to participate in vaccine or antiviral therapy trials, and 2) allow for ready procurement of biological specimens from healthy volunteers to facilitate rapid research assay development.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age: 18 or older
* Available to participate for the planned duration of at least one clinical trial for which screening is being done or to donate blood, nasal swab, throat swab, and/or urine in support of assay development
* Able and willing to complete the informed consent process
* Agree to have blood and/or urine, stool, nasal swab, or wash samples collected as needed for the clinical trial screening or sample donation process
* Agree to participate in procedures, such as electrocardiogram or pulmonary function tests, as may be needed for the clinical trial screening process
* Do not have plans to become pregnant while on this study
* Able to provide a medical history and other relevant personal information as appropriate

EXCLUSION CRITERIA:

* A condition that requires active medical intervention or monitoring to avert serious danger to the participant s health or well-being
* Known to be pregnant or breast-feeding
* If planning to enroll in a clinical trial, the receipt of immunoglobulin within the past 6 months or anticipated within the next year
* Any other condition that in the opinion of the investigator would make the subject unsuitable for enrollment or could interfere with the subject participating in and completing the study or a specimen donation.
* Use of recreational drugs or alcohol dependency or abuse

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers, male or female ages 18-65.@@@
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
To develop a pool of subject eligible to participate in clinical trials of investigational or licensed vaccines or antiviral products. | Within one year from enrollment of each individual.
  A pool of subjects qualified to participate in clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Davey, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-I-0194.html